CLINICAL TRIAL: NCT04000841
Title: Culturally Responsive Stress Reduction: A Mobile Mindfulness Application to Support Health Promotion for African Americans
Brief Title: Culturally Responsive Stress Reduction: A Mobile Mindfulness Application for African Americans (CRSR)
Acronym: CRSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRIS Media Inc (Other)
Collaborators: Spelman College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2R44MD012284-02 (NIH)
Record Dates: First submitted 2019-06-20; First posted 2019-06-27 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Behavior
Keywords: stress; emotion regulation
MeSH Terms: conditions — Behavior; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention participants receive access to the Mindful You app for 12 weeks. They will use the app to listen to guided meditations and to receive notifications, messages, and reminders that they select and ones sent to all participants by the app.
  Interventions: Behavioral: Mindful You mobile app
- Waitlist Control (No Intervention): Waitlist control participants will continue business as usual with regards to stress-management and reduction.

INTERVENTIONS:
Behavioral: Mindful You mobile app — The CRSR intervention consists of a native mobile application for Android and iOS devices. The mobile app includes:
  * Guided meditations of varying length designed to connect the user to the present moment and a place of calm through culturally aligned exercises grounded in spirituality, orality, self-empowerment, and resilience.
  * User-customized notifications prompting users to reflect and engage with the app, such as providing African American proverbs and quotes and asking simple questions like "What are you grateful for today?"
  * Scheduled messages on the importance mindfulness as a way increase control over physical and psychological health
  * User-customized reminders to do specific meditations and display personally selected images or messages.
  Arms: Intervention

SUMMARY:
Over a 12-week period the investigators will test whether, compared to the Waitlist-Control (WC) condition, administration of the full CRSR intervention improves participants self-reported outcomes of stress, self-efficacy, mindfulness, use of mindfulness strategies, and knowledge. The investigators also will examine the usability, cultural relevance, and user satisfaction.

DETAILED DESCRIPTION:
The proposed intervention, Culturally Responsible Stress Reduction: A Mobile Mindfulness Application to Support Health Promotion for African Americans (CRSR), is designed to encourage the use of mindfulness to mitigate the disproportionate amount of stress-related health disparities facing African Americans. Current mindfulness approaches have been unsuccessful in engaging this population. This proposal aims to bridge this disparity by developing an mHealth (mobile health) mindfulness application ("app") tailored specifically to the cultural values of the African American community.

Mindfulness involves meditative practices that cultivate purposeful and nonjudgmental attention to current thoughts, emotions, and physical sensations in the body. Mindfulness has been incorporated into widely-used interventions, including Acceptance and Commitment Therapy (ACT). The CRSR app will be grounded in ACT and will integrate the convenience of mobile technology with tailored content to allow users to shift from potentially harmful culturally prescribed stress-coping activities (e.g., self-reliance, emotional suppression) to adaptive mindfulness-based stress-coping activities aligned with culturally specific values. This integration of content, backed by theory and empirical evidence, effective instructional delivery, an interdisciplinary development team, and modern communication technology will produce an effective mHealth intervention.

The CRSR app features include guided meditations to connect the user to the present moment and a place of calm through culturally aligned exercises grounded in spirituality, orality, self-empowerment, and resilience; personalized notifications prompting users to reflect and engage with the app; periodic email messages on the importance mindfulness as a way increase control over physical and psychological health; and user-customized reminders.

Phase I included developing a testable prototype of the CRSR app, called Mindful You. The prototype provided functionality for participants to practice mindfulness and was used to test proof of concept, i.e., the feasibility and social acceptability of the CRSR app. Users experienced significantly decreased stress and increased self-efficacy. They also reported increased use of mindfulness behaviors and improved self-regulation. Phase II will iteratively build on the prototype to develop the final product and test its efficacy with a fully-powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as African-American
* Can read, write, and understand English
* Have a valid email address
* Owns an iOS or Android mobile device

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress | Baseline and 12 weeks
  Stress will be assessed using the Perceived Stress Scale (PSS), a 10-item frequency scale that evaluates the amount of stress in one's life.Scale ranges from 1 (never) to 4 (very often) with higher scores indicating more stress, therefore decreases at posttest would indicate better outcomes. The scores are averaged to get a total score on the scale which has good internal reliability (alpha = .90 in Phase I).

SECONDARY OUTCOMES:
Change in Emotion Regulation | Baseline and 12 weeks
  Emotion regulation will be assessed by the Difficulty in Emotion Regulation Scale Short Form (DERS-SF), a 18 item frequency scale ranging from 1 (almost never; 0-10%) to 5 (almost always; 91-100%) with higher scores indicating less emotional regulation (negative change scores indicate better outcomes). Single score and 6 subscales (strategies, non-acceptance, impulse, goals, awareness, and clarity) can be analyzed as either total score or average scores. Total scores on the full scale range from 18 to 90. Subscales have three items each, thus total scores on the subscales range from 3 to 15.
Change in Mindfulness | Baseline and 12 weeks
  Mindfulness will be assessed by the Five Facet Mindfulness Questionnaire (FFMQ), a 24-item frequency scale with scores ranging from 1 (never) to 5 (very often). This scale provides subscales with four having five items each (describe, act with awareness, nonjudgmental, and non-reactance) and on having four items (observe). Total scores range from 5 to 25 on the five-item subscales and 4 to 20 on the four-item subscale, with higher scores indicating indicating more mindfulness. Thus positive changes at posttest indicate better outcomes.
Change in Attitudes toward Mindfulness | Baseline and 12 weeks
  Attitudes toward general use of mindfulness techniques as well as program specific recommendations, affective responses towards the items, and outcome expectancies will be measured using the Attitudes Towards Mindfulness Scale (MTMS), a 10-item scale developed in Phase I. The MTMS is a 10-item Likert-like scale, on a 5 point scale ranging from 1 "strongly disagree" to 5 "strongly agree" which measured positive attitudes towards mindfulness strategies (higher change scores indicate a better outcome). Example items included "Practicing mindfulness can help me reduce my stress" and "Knowing what I am thinking in the moment is important". The MTMS demonstrated strong internal reliability during Phase I (alpha = .91 at pretest and .94 at posttest). The average score of the scale is used in analysis.
Change in Perceived Behavioral Control | Baseline and 12 weeks
  Perceived Behavioral Control (self-efficacy) will be measured using the Mindfulness Self-Efficacy Scale (MSES) a 12-item Likert-like scale developed in Phase I based on the content about ability and competence in stress reduction through mindfulness. The MSES evaluated self-efficacy, by asking how confident on a 5 point scale ranging from 1 "not at all confident" to 5 "very confident" participants were in their ability to use the skills taught in the course, for example "Take time to breathe" and "Pay attention to tasks in the moment". Higher scores indicated greater self-efficacy (better outcome). The MSES demonstrated strong internal reliability in Phase I (alpha = .90 at pretest and .91 at posttest). The average score of the scale is used in analysis.
Change in Mindfulness Behaviors | Baseline and 12 weeks
  Mindfulness Behaviors i.e., actual behavioral change, will be assessed through the Mindfulness Behavior Usage Scale (MBUS) a self-report of 12 mindfulness activities as well as usage data provided through the app. The MBUS is a 12-item frequency scale, asking how often in the last week participants engaged in mindfulness strategies, ranging from 1 "never' to 4 "daily" (higher change scores indicate better outcomes). For example, "How often did you take time to breathe" and "Pay attention to tasks in the moment". The MBUS demonstrated good internal reliability (alpha = .94 at pretest and .90 at posttest).
Change in Knowledge of Mindfulness | Baseline and 12 weeks
  Knowledge about mindfulness techniques will be assessed pre- and post- to determine the extent to which participants understand basic knowledge delivered during the intervention. Knowledge items will be derived from the conceptual and practical content. In Phase I we used a 10-item multiple-choice assessment of participants' knowledge about mindfulness. For Phase II additional items will be added to reflect the new information presented in the program.

CONTACTS AND LOCATIONS:
Locations (1):
- IRIS Educational Media, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No